CLINICAL TRIAL: NCT04133441
Title: 25-Hydroxyvitamin D Levels Are Negatively Associated With Platelets Number in a Cohort of Overweight and Obese Subjects
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: vitDplatelet
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was aimed to investigate the associations between platelet number and 25(OH)D serum concentration in apparently healthy but overweight/obese subjects.

DETAILED DESCRIPTION:
Subjects were enrolled at the first examination whether they were not taking any medication, including oral contraceptives or drugs for osteoporosis, and free of significant medical illnesses, except obesity. Exclusion criteria were history of endocrinological diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.), chronic inflammatory diseases, stable known hypertension, angina pectoris, stroke, transient ischemic attack, heart infarction, congenital heart disease, malignancies, chronic inflammatory diseases, renal and liver failure, angina pectoris, myocardial infarction, heart failure, congenital heart diseases, minor and major stroke, and inherited thrombocytopenias and other major malignancies. subjects were examined by means of the medical history, hormonal, metabolic and routine hematochemical parameters. We provided for a clinical baseline evaluation that included extemporaneous ambulatory blood pressure (BP) and a physical assessment of body weight, Body Mass Index (BMI) and Waist Circumference (WC) as anthropometric parameters. To lead the statistical analysis, all sample was clusterized into three different groups according to the diagnostic condition of deficiency (<10 ng/mL), insufficiency (<20 ng/mL) and sufficiency (≥20 ng/mL) of vitamin D. We labelled each cluster as group 1, group 2 and group 3.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI> 25 Kg/m2)

Exclusion Criteria:

* Any kind of drug
* Hypertension
* Endocrine diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.),
* Chronic inflammatory diseases
* Renal failure
* Liver failure
* Angina pectoris
* Myocardial infarction and heart failure
* Genetic heart diseases
* Thrombocytopenias

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who came to the Outpatient Clinic of Nutrition at the National Institute of Gastroenterology "S. de Bellis," Research Hospital, Castellana Grotte, Italy.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D | At baseline
  Vitamin D (ng/mL) concentration in serum
Platelets | At baseline
  Platelets (cells/mm3) number in serum

SECONDARY OUTCOMES:
Insulin | At baseline
  Insulin (mIU/L) concentration in serum
eGFR (estimated glomerular filtration rate) | At baseline
  eGFR (ml/min/1.73 mq)
Creatinin | At baseline
  Creatinin (mg/dl) concentration in serum
Total cholesterol | At baseline
  Total cholesterol (mg/dL) concentrations in serum
Thyroid hormones (FT3, FT4) | At baseline
  FT3 (pg/mL), FT4 (pg/mL) concentration in serum
HDL cholesterol | At baseline
  HDL cholesterol (mg/dL) concentrations in serum
LDL cholesterol | At baseline
  LDL cholesterol (mg/dL) concentrations in serum
TSH | At baseline
  TSH (mU/L) concentration in serum
BMI | At baseline
  BMI (kg/m^2)
Height | At baseline
  Height in meters
Weight | At baseline
  Weight in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Gastroenterology IRCCS S. de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No